CLINICAL TRIAL: NCT06751732
Title: Effects of Craniocervical Flexion Training on Headache Frequency, Intensity, and Functional Disability in Patients With Migraine
Brief Title: Craniocervical Flexion Training for Reducing Migraine Headaches and Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Muhammad Husnain
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Episodic Migraine Headache
Keywords: Migraine; Non-Pharmacological Interventions; Physiotherapy; Craniocervical Flexion Training; Craniocervical Flexion Exercises
MeSH Terms: conditions — Migraine Disorders | interventions — Traction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Comprehensive Physiotherapy Protocol with Craniocervical Flexion Training (CCFT) (Experimental): The physiotherapy protocol will consist of the following components:
  Diaphragm Respiratory Training (15 minutes), Cervical Mobilization and Traction (5 minutes), Digital Compression on Muscle Trigger Points (6 minutes), Passive Stretching of Neck Muscles, Passive Stretching of Neck Muscles, Instruction on Postural Correction and Specialized Craniocervical Flexion Training (CCFT) Protocol.
  Interventions: Other: Craniocervical Flexion Training (CCFT); Other: Diaphragm Respiratory Training; Other: Cervical Mobilization and Traction; Other: Digital Compression on Muscle Trigger Points; Other: Passive Stretching of Neck Muscles; Other: Instruction on Postural Correction
- Group B: Comprehensive Physiotherapy Protocol without Craniocervical Flexion Training (CCFT) (Active Comparator): Participants in Group B will receive the same comprehensive physiotherapy protocol as Group A, excluding the specialized CCFT.
  Interventions: Other: Diaphragm Respiratory Training; Other: Cervical Mobilization and Traction; Other: Digital Compression on Muscle Trigger Points; Other: Passive Stretching of Neck Muscles; Other: Instruction on Postural Correction

INTERVENTIONS:
Other: Craniocervical Flexion Training (CCFT) — CCFT is a targeted intervention aimed at improving neuromuscular control in the cervicoscapular and craniocervical regions through low-load endurance exercises. A pressure biofeedback unit placed behind the neck sets a baseline at 20 mmHg, ensuring relaxed neck muscles. Participants open the mouth 20 mm to activate deep cervical flexors and minimize superficial muscle use, maintaining head contact with the surface while gazing 45 degrees below the horizontal. Pressure is increased in 5 mmHg steps (20 to 40 mmHg), with each level held for 10 seconds, followed by a 10-second rest. CCFT can also be performed seated, reducing sternocleidomastoid activity and promoting longus colli thickness for functional training.
  Arms: Group A: Comprehensive Physiotherapy Protocol with Craniocervical Flexion Training (CCFT)
Other: Diaphragm Respiratory Training — Patients will undergo a 15-minute diaphragmatic respiratory training session, focusing on smooth diaphragmatic breathing with gentle expirations.
Other: Cervical Mobilization and Traction — A physiotherapist will perform a low-velocity, passive cervical joint mobilization technique (Oscillation technique) based on the regimen described by Maitland.(17) This will be followed by cervical spine traction while patients continue diaphragmatic breathing.
Other: Digital Compression on Muscle Trigger Points — Digital compression will be applied for 90 seconds on identified trigger points in the craniocervical muscles, not exceeding eight trigger points in each session.
Other: Passive Stretching of Neck Muscles — Passive stretching will be performed three times for neck flexion and rotation associated with ipsilateral flexion directions, using moderate force within the patient's pain limits, and maintained for 30 seconds.
Other: Instruction on Postural Correction — Physiotherapists will provide instructions on postural correction, addressing craniocervical extension, cervicothoracic flexion, protraction of shoulders, increased thoracic kyphosis, and flattened lumbar lordosis. Patients will be guided on correcting these postural abnormalities through craniocervical flexion, cervicothoracic extension, shoulder retraction, thoracic spine extension, and normalization of lumbar lordosis.

SUMMARY:
Migraine, a leading cause of disability globally, necessitates effective interventions beyond pharmacotherapy due to the associated risks. This project addresses the literature gap by focusing on physiotherapy, particularly novel craniocervical flexion training (CCFT), for managing migraine headache. The prevalence of migraines, coupled with their economic burden, underscores the urgency for non-pharmacological alternatives. Current pharmacological treatments pose challenges, making nonpharmacological modalities like exercise physiotherapy and manual therapy promising migraine management. Despite limited research, these interventions show potential benefits in addressing peri-cranial muscle tenderness and cervical dysfunction. This study aims to assess the effects of a comprehensive physiotherapy protocol, including the CCFT, shedding light on its impact on migraine frequency, onset, and intensity.

This Randomized Clinical Trial will be conducted at Riphah Rehab Training and Research Center, spans 8 months. The sample size of 38 individuals will undergo a comprehensive physiotherapy protocol, either with or without the CCFT. Data collection, occurring at baseline, 2 weeks, and 4 weeks, includes primary outcomes (headache frequency, intensity, HIT-6 scores) and secondary outcomes (MSQ. V2.1). Participants will receive a minimum of 2 sessions per week, maintaining confidentiality. Randomization, conducted by computer-generated stratified randomization, ensures unbiased allocation to the two groups. The single-blind study incorporates rigorous statistical analysis, utilizing SPSS software for descriptive statistics, change over time assessments, and intergroup differences via t-tests and f-tests.

DETAILED DESCRIPTION:
Migraine along with tension-type headache and cluster-headache are three major types of primary headaches. Through the Global Burden of Disease (GBD) study, headache disorders are revealed as one of the major public-health concerns globally in all countries and world regions. In the 2019 iteration (GBD2019), migraine alone was second among the causes of disability, and first among women under 50 years of age. The data indicated that the worldwide prevalence of migraine was approximately 14.0% (8.6% in males, 17.0% in females), while tension-type headache (TTH) had a prevalence of 26.0% (23.4% in males, 27.1% in females). The International Classification of Headache Disorders version 3 (ICHD-3) defines primary headache as a headache disorder not caused by or attributed to another disorder. Primary headaches are disorders by themselves. They are caused by independent Patho-mechanisms and not by other disorders. Using economic loss due to migraine and working population data from the Statistics Bureau of Japan, the annual economic loss due to presenteeism is US $3.3 billion, calculated from the number of days when work efficiency has fallen to less than half due to headaches using Migraine Disability Assessment Questionnaire (MIDAS).

The pharmacological approach is one of the first-line treatments within the international guidelines for treating primary headaches. The main classes of drugs to treat migraine headaches include: Beta-blockers, Anticonvulsants, Antidepressants, and other prophylactic medications. Medication overuse cause a significant bad effect to those with primary headaches, potentially leading to a shift from episodic headache attacks to chronic headache episodes. Therefore, guidelines already implement nonpharmacological modalities in the management of primary headaches as main treatments within the physical therapy practice. Manual Therapy is one of the most common nonpharmacological treatments used for the management of common recurrent headaches.

Limited research exists on physical therapy for treating migraines, but it can still offer benefits. Migraine sufferers may experience tender peri-cranial muscles and altered muscle tone and cervical dysfunction between episodes. Physical therapy interventions, including manual therapy, targeted exercises, education, and modalities, can help reduce attack frequency, onset, and intensity. There are many MT interventions available for headache disorders which are mostly applied on cervical region. A study on the treatment of neck pain for migraine patients showed better response to physiotherapy as compared to aerobic exercises.

The prevalence of migraines globally, as indicated by the Global Burden of Disease study, underscores the urgent need for effective interventions. Migraine not only ranks among the leading causes of disability but also imposes a substantial economic burden. Current pharmacological approaches, while commonly employed, carry the risk of medication overuse and the transition from episodic to chronic headaches. Recognizing the limitations of pharmacotherapy, nonpharmacological modalities, particularly exercise physiotherapy and manual therapy (MT), emerge as promising avenues for managing migraines. Although research on physical therapy for migraines is limited, its potential benefits, such as addressing peri-cranial muscle tenderness and cervical dysfunction, make it a valuable area of exploration. This research seeks to evaluate the efficacy of a novel CCFT am within the context of manual therapy, providing insights into its impact on migraine frequency, onset, and intensity.

ELIGIBILITY:
Inclusion Criteria:

• Patients diagnosed with episodic Migraine. A diagnosis of episodic migraine will be made by the primary investigator under the guidance of a medical practitioner as per the ICHD-3. An episodic migraine is that which occurs on less than 15 days per month for at least 3 months.(4)

Exclusion Criteria:

* Headache diagnosis: Other than migraine according to ICHD-3
* Upper cervical spine instability.(21)
* Cervical arterial insufficiency.
* Vertigo or dizziness history.
* Rheumatoid arthritis, ankylosing spondylosis, cervical spine fractures.
* Pregnancy.
* Cognitive compromise.
* Contraindications to manual therapy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | baseline, after 4 weeks, and after 3 months
  The Numeric Pain Rating Scale (NPRS) is a pain assessment tool where patients rate their current pain intensity on an 11-point numeric scale, ranging from 0 ("absence of pain") to 10 ("most severe pain imaginable"). While the Minimal Clinically Important Difference (MCID) is established as 1.3 in individuals with mechanical neck pain12, this specific value hasn't been documented for patients with cervical radiculopathy (CR). Recent findings indicate moderate test-retest reliability (ICC = 0.63) in individuals with CR.
The Migraine Disability Assessment Test | baseline, after 4 weeks, and after 3 months
  The Migraine Disability Assessment Test (MIDAS) is a widely used, standardized tool designed to measure the impact of migraines on an individual's daily life. It assesses the degree of disability caused by migraines over the previous three months, focusing on areas such as work, household activities, and social or leisure engagements. The test consists of five key questions addressing the number of days migraines affected productivity or routine activities, along with an additional question on headache frequency. Scores are categorized into disability levels, ranging from minimal to severe, to guide clinical decisions and treatment planning.
A headache diary | baseline, after 4 weeks, and after 3 months
  A headache diary by the national headache foundation will be used to keep track of the headache episodes, intensity, and other parameters.

SECONDARY OUTCOMES:
Headache Impact Test questionnaire (HIT-6) | baseline, after 4 weeks, and after 3 months
  The Head Impact Test (HIT-6) exhibited high internal consistency reliability (0.82-0.90) and test-retest reliability (0.77) among migraine sufferers. Construct validity was supported by correlations with Migraine Disability Assessment Questionnaire (MIDAS) and negative correlations with SF-8 scales. Discriminant validity was observed across headache stages. Score for HIT-6 ranges from 36 to 78. Greater score means greater impact on life. The HIT-6's smaller difference between chronic and episodic migraine scores (2.3) compared to MIDAS (21.6) underscores its effectiveness in evaluating subjective impact. Both instruments assess different aspects of headache-related disability. The HIT-6's one-month recall offers a more accurate evaluation than the MIDAS's three-month recall.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Husnain Irshad, DPT, Principal Investigator — Riphah International University, Lahore; Syed Shakil ur Rehman, PhD, Study Director — Riphah International University, Lahore
Locations (1):
- Riphah Rehab Training and Research Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No